CLINICAL TRIAL: NCT04505540
Title: Effectiveness of Bridge Clinic Following Emergency Department-Initiated Intervention for Opioid Use Disorder
Brief Title: Start Treatment and Recovery for Opioid Use Disorder
Acronym: STAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vermont (Other)
Collaborators: Substance Abuse and Mental Health Services Administration (SAMHSA) (U.S. Federal Agency); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Scott Mackey, Assistant Professor, University of Vermont
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CHRMS: 18-0695; 1R21DA049859-01 (NIH)
Record Dates: First submitted 2020-06-11; First posted 2020-08-10 (Actual); Results first posted 2023-12-11 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Opioid-use Disorder; Mental Disorder; Opioid Medication Assisted Treatment
MeSH Terms: conditions — Opioid-Related Disorders; Mental Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Bridge Clinic (Experimental): Medication assisted treatment supervised by addiction bridge clinic until stabilized in treatment.
  Interventions: Other: Bridge Clinic

INTERVENTIONS:
Other: Bridge Clinic — Specialized addiction bridge clinic

SUMMARY:
The purpose of this study is 1) to evaluate whether emergency department-initiated medically assisted treatment with Buprenorphine/Naloxone in patients presenting with opioid use disorder will produce positive outcomes at 1 week, 3 months and 6 months after treatment initiation.

DETAILED DESCRIPTION:
The emergency department is a critical missed opportunity to engage patients with opioid use disorder in medication-assisted treatment, the most effective current treatment for the disorder. Patients presenting at the emergency department with opioid use disorder will be given the opportunity to immediately start medication assisted treatment with Naloxone/Buprenorphine then referred either to a specialized addiction bridge clinic or a local waivered provider for further treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patient at Emergency Department
* Diagnosis opioid use disorder according to criteria Diagnostic and Statistical Manual (DSM) 5

Exclusion Criteria:

* Participating in alternate treatment program for opioid use disorder
* Prisoner
* Inability to communicate
* Psychosis
* Suicidality
* History of Buprenorphine injection
* Critical Illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2019-09-30 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-10-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Vermont Medical Center, Burlington, Vermont, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Baseline
Arm/Group | Bridge Clinic
Started | 104
Completed | 94
Not Completed | 10
Not completed — Protocol Violation | 10
Period: 1 Week Eligible to Self-report
Arm/Group | Bridge Clinic
Started | 94
Completed | 93
Not Completed | 1
Not completed — Incarcerated/Institutionalized | 1
Period: 1 Week Contacted for Self-report
Arm/Group | Bridge Clinic
Started | 93
Completed | 66
Not Completed | 27
Not completed — Lost to Follow-up | 27
Period: 1 Week Eligible for Urinanalysis
Arm/Group | Bridge Clinic
Started | 94 (Self-reports on treatment retention and urine sampling were conducted separately.)
Completed | 41
Not Completed | 53
Not completed — COVID disruption of urine sampling | 52
Not completed — Incarcerated/Institutionalized | 1
Period: 1 Week Urine Sample Provided
Arm/Group | Bridge Clinic
Started | 41
Completed | 28
Not Completed | 13
Not completed — Lost to Follow-up | 13
Period: 3 Months Eligible to Self-report
Arm/Group | Bridge Clinic
Started | 94 (Note the protocol followed an intent-to-treat protocol. Participants who were eligible but did not complete a questionnaire or urinalysis were counted as negative for enrollment in treatment and positive for illicit drug use. Participants were not withdrawn if they did not complete 1 week or 3 months testing and were considered eligible again for contact at the next stage.)
Completed | 87
Not Completed | 7
Not completed — Incarcerated/Institutionalized | 7
Period: 3 Months Contacted for Self-report
Arm/Group | Bridge Clinic
Started | 87
Completed | 65
Not Completed | 22
Not completed — Lost to Follow-up | 22
Period: 3 Months Eligible for Urinanalysis
Arm/Group | Bridge Clinic
Started | 94 (Note the protocol followed an intent-to-treat protocol. Participants who were eligible but did not complete a questionnaire or urinalysis were counted as negative for enrollment in treatment and positive for illicit drug use. Participants were not withdrawn if they did not complete 1 week or 3 months testing and were considered eligible again for contact at the next stage.)
Completed | 24
Not Completed | 70
Not completed — COVID disruption of urine sampling | 70
Period: 3 Months Urine Sample Provided
Arm/Group | Bridge Clinic
Started | 24
Completed | 11
Not Completed | 13
Not completed — Lost to Follow-up | 13
Period: 6 Months Eligible to Self-report
Arm/Group | Bridge Clinic
Started | 94 (Note the protocol followed an intent-to-treat protocol. Participants who were eligible but did not complete a questionnaire or urinalysis were counted as negative for enrollment in treatment and positive for illicit drug use. Participants were not withdrawn if they did not complete 1 week or 3 months testing and were considered eligible again for contact at the next stage.)
Completed | 85
Not Completed | 9
Not completed — Incarcerated/Institutionalized | 9
Period: 6 Months Contacted for Self-report
Arm/Group | Bridge Clinic
Started | 85
Completed | 68
Not Completed | 17
Not completed — Lost to Follow-up | 17
Period: 6 Months Eligible for Urinanalysis
Arm/Group | Bridge Clinic
Started | 94 (Note the protocol followed an intent-to-treat protocol. Participants who were eligible but did not complete a questionnaire or urinalysis were counted as negative for enrollment in treatment and positive for illicit drug use. Participants were not withdrawn if they did not complete 1 week or 3 months testing and were considered eligible again for contact at the next stage.)
Completed | 3
Not Completed | 91
Not completed — COVID disruption of urine sampling | 91
Period: 6 Months Urine Sample Provided
Arm/Group | Bridge Clinic
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: 94 participants were available for analysis after 10 were withdrawn from the study
Arm/Group | Bridge Clinic
Number analyzed (Participants) | 94
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.6 (8.7)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male/Female/Unknown: Male | 60
  Male/Female/Unknown: Female | 33
  Male/Female/Unknown: Unknown | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 77
  More than one race | 4
  Unknown or Not Reported | 9
Region of Enrollment [Number; unit: participants]
  United States | 94

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Self-reported Treatment Retention
Description: Self-reported enrollment in treatment for opioid use disorder after 1 week
Time Frame: 1 week
Measure: Count of Participants; unit: Participants
Arm/Group | Bridge Clinic
Number analyzed (Participants) | 93
Participants | 51

2. Primary Outcome: Number of Participants With Self-reported Treatment Retention
Description: Self-reported enrollment in treatment for opioid use disorder after 3 months
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Bridge Clinic
Number analyzed (Participants) | 87
Participants | 49

3. Primary Outcome: Number of Participants With Self-reported Treatment Retention
Description: Self-reported enrollment in treatment for opioid use disorder after 6 months
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Bridge Clinic
Number analyzed (Participants) | 85
Participants | 51

4. Secondary Outcome: Number of Participants With Illicit Opioid Use
Description: Urine analyzed for opioids (buprenorphine, methadone, oxycodone, hydrocodone, hydromorphone, heroin, fentanyl) and other drugs (cocaine, amphetamines, benzodiazepines, cannabinoids) via enzyme multiplied immunoassay. Note buprenorphine and methadone positive results not treated as illicit.
Time Frame: 1 week
Measure: Count of Participants; unit: Participants
Arm/Group | Bridge Clinic
Number analyzed (Participants) | 41
Participants | 20

5. Secondary Outcome: Number of Participants With Illicit Opioid Use
Description: as for outcome 4
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Bridge Clinic
Number analyzed (Participants) | 24
Participants | 14

6. Secondary Outcome: Number of Participants With Illicit Opioid Use
Description: as for outcome 4
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Bridge Clinic
Number analyzed (Participants) | 3
Participants | 1

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Bridge Clinic
All-Cause Mortality (participants affected / at risk) | 0/94
Serious Adverse Events (participants affected / at risk) | 0/94
Other Adverse Events (participants affected / at risk) | 0/94

LIMITATIONS AND CAVEATS:
Urinalysis was disrupted by the COVID-19 epidemic. Consequently, urinalysis at 1 week, 3 months, and 6 months (although reported) should be regarded with caution.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-07): https://cdn.clinicaltrials.gov/large-docs/40/NCT04505540/Prot_SAP_000.pdf